CLINICAL TRIAL: NCT02342236
Title: The Regional Cerebral Oxygen Saturation and Both S100B and GFAP Proteins Serum Concentration in Patients Undergoing Primary Hip Arthroplasty.
Brief Title: Cerebral Regional Oxygen Saturation and Markers of Brain Damage During Primary Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Dariusz Tomaszewski, M.D., Ph.D., Military Institute od Medicine National Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 06101968-3
Record Dates: First submitted 2015-01-05; First posted 2015-01-19 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Delirium, Dementia, Amnestic, Cognitive Disorders; Arthroplasty, Hip Replacement
Keywords: Biological Markers
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- cemented (Other): Primary hip arthroplasty with bone cement use.
  Interventions: Device: cemented or cementless type of hip prothesis
- cementless (Other): Primary hip arthroplasty without bone cement use.
  Interventions: Device: cemented or cementless type of hip prothesis

INTERVENTIONS:
Device: cemented or cementless type of hip prothesis

SUMMARY:
Postoperative Cognitive Disorders (POCD) are common in hospitalized people > 60 year old, especially in orthopedic patients. Etiology of POCD is complex, and in some aspects still remains unclear. The role of thromboembolic events in etiology of POCD was discussed. The incidence of such events in patients who underwent big joints arthroplasty can be as high as 40 to 60%, although some cases are subclinical. Thromboembolic material can block a blood flow through a vessels in the brain. As a consequence cerebral neurons can be damaged or destroyed. After neuronal damage specific substances, such as S100B protein, glial fibrillary acidic protein (GFAP) and neuron-specific enolase (NSE) are released to the blood. The serum concentrations of these biomarkers can be measured. Moreover, the block of blood flow will decrease regional cerebral saturation in affected parts of the brain.

In this project the authors would like to analyze the correlation between the regional cerebral saturation and serum concentration of both S100B protein and GFAP in orthopedic patients scheduled to primary hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled to primary hip arthroplasty,
* orthopedic procedure under spinal anesthesia.

Exclusion Criteria:

* patients younger than 18 y.o.,
* surgery under general anesthesia,
* patients who refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in regional cerebral oxygen during primary hip arthroplasty | Duration of the orthopedic procedure, an expected average of 2 hours.
  The analysis of regional cerebral oxygen saturation will start just before the anesthesia and ends just after the surgery.

SECONDARY OUTCOMES:
Changes in serum levels of S100B protein from baseline at 72 hours after the surgery | 72 hours
  The serum concentration of S100B protein will be measured [1] just before the surgery, [2] just after the end of the surgery, an expected average of two hours, [3] 6 hours after the beginning of the surgery, [4] 24 hours after the beginning of the surgery, and [5] 72 hours after the beginning of the surgery.
Changes in serum levels of GFAP from baseline at 72 hours after the surgery | 72 hours
  The serum concentration of GFAP protein will be measured [1] just before the surgery, [2] just after the end of the surgery, an expected average of two hours, [3] 6 hours after the beginning of the surgery, [4] 24 hours after the beginning of the surgery, and [5] 72 hours after the beginning of the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Therapy, Warsaw, Poland

REFERENCES:
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Background] Colonna DM, Kilgus D, Brown W, Challa V, Stump DA, Moody DM. Acute brain fat embolization occurring after total hip arthroplasty in the absence of a patent foramen ovale. Anesthesiology. 2002 Apr;96(4):1027-9. doi: 10.1097/00000542-200204000-00036. No abstract available. PMID 11964616
- [Background] Vos PE, Jacobs B, Andriessen TM, Lamers KJ, Borm GF, Beems T, Edwards M, Rosmalen CF, Vissers JL. GFAP and S100B are biomarkers of traumatic brain injury: an observational cohort study. Neurology. 2010 Nov 16;75(20):1786-93. doi: 10.1212/WNL.0b013e3181fd62d2. PMID 21079180
- [Background] Nylen K, Csajbok LZ, Ost M, Rashid A, Blennow K, Nellgard B, Rosengren L. Serum glial fibrillary acidic protein is related to focal brain injury and outcome after aneurysmal subarachnoid hemorrhage. Stroke. 2007 May;38(5):1489-94. doi: 10.1161/STROKEAHA.106.478362. Epub 2007 Mar 29. PMID 17395862
- [Background] Wiesmann M, Steinmeier E, Magerkurth O, Linn J, Gottmann D, Missler U. Outcome prediction in traumatic brain injury: comparison of neurological status, CT findings, and blood levels of S100B and GFAP. Acta Neurol Scand. 2010 Mar;121(3):178-85. doi: 10.1111/j.1600-0404.2009.01196.x. Epub 2009 Oct 5. PMID 19804476
- [Background] Slater JP, Guarino T, Stack J, Vinod K, Bustami RT, Brown JM 3rd, Rodriguez AL, Magovern CJ, Zaubler T, Freundlich K, Parr GV. Cerebral oxygen desaturation predicts cognitive decline and longer hospital stay after cardiac surgery. Ann Thorac Surg. 2009 Jan;87(1):36-44; discussion 44-5. doi: 10.1016/j.athoracsur.2008.08.070. PMID 19101265